CLINICAL TRIAL: NCT05645328
Title: Effectiveness and Implementation of a Health System Intervention to Improve Quality of Cancer Care for Rural, Underserved Patients
Brief Title: Implementation of a Health System Intervention to Improve Quality of Cancer Care for Rural Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Charlton (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mary Charlton, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 202202104; R01CA254628 (NIH)
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Health system intervention; Rural health; Quality improvement; Implementation science
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Hospital Administrators, Providers, and Data Monitoring Staff (Experimental): This is a health-system-level intervention, designed as two-arm intervention trial, where four participating hospitals will be offered support in the areas of training and education, cancer data collection and reporting, quality improvement and clinical peer-to-peer support.
  Hospitals that are eligible for the intervention had to be located in an Iowa county classified as non-metropolitan according to rural urban continuum codes (RUCC) 4 through 9 and diagnose or treat at least 100 cancer patients each year. We selected 4 of the 9 rural hospitals meeting this criteria to administer the intervention.
  Interventions: Other: Iowa Cancer Affiliate Network (ICAN)
- Control arm (No Intervention): Hospitals that are eligible for the intervention had to be located in an Iowa county classified as non-metropolitan according to rural urban continuum codes (RUCC) 4 through 9 and diagnose or treat at least 100 cancer patients each year. The remaining 5 hospitals meeting this criteria that were not selected for the intervention will serve as controls.

INTERVENTIONS:
Other: Iowa Cancer Affiliate Network (ICAN) — Each hospital in the intervention has undergone interviews in which the investigators elicited program goals, challenges, and readiness for change. Prior to the intervention, the cancer centers will be provided a document specifying current status for meeting Commission on Cancer (CoC) accreditation standards, gaps identified, suggestions and resources for the next steps to meet goals, and progress toward fulfilling CoC accreditation standards. The hospitals will be offered support, expertise, and resources to facilitate them in achieving the CoC standards. Support will be offered in the form of education/training regarding the standards and provision of cancer services, regular in-person/zoom check-ins with hospital stakeholders to evaluate progress, and provision of documentation/educational resources regarding standard requirements. The intervention actions will be tailored to the needs of each hospital based on standards they currently do not meet and choose to work toward.
  Arms: Intervention Hospital Administrators, Providers, and Data Monitoring Staff

SUMMARY:
The purpose of this study is to implement and evaluate the recently developed Iowa Cancer Affiliate Network (ICAN) intervention.

The ICAN intervention will consist of members of the research team providing ongoing support to participating hospitals in achieving the quality standards outlined by the American College of Surgeons Commission on Cancer (CoC). Support will be offered in the form of education and training regarding the standards and provision of cancer services, regular in-person and zoom check-ins with hospital stakeholders to evaluate progress, and provision of documentation and educational resources regarding standard requirements.

Implementation approach:1) Engage implementation teams and develop and execute implementation plans based on hospital needs assessments; and 2) Conduct interviews with key ICAN stakeholders to assess acceptability, adoption, appropriateness and cost (based on Proctor's implementation outcomes framework) and determinants of these outcomes (e.g., hospital structure, culture, resources, capacity, readiness) based on the Consolidated Framework for Implementation Research.

Evaluation approach: Using Iowa Cancer Registry data routinely collected for surveillance purposes, the investigators will compare rates of compliance with pre- and post-intervention treatment-related quality measures in target and control hospitals. The rural hospitals in Iowa that serve the most rural cancer patients and have never been accredited by the CoC were chosen for intervention targets, and all committed to participating in the study (letters of support provided). The remainder of rural hospitals that care for >100 newly diagnosed cancer patients per year (n=5) were chosen as a comparison group. The investigators will use data routinely collected by the Iowa Cancer Registry to compare aggregate compliance with quality measures for cancer care between the hospitals included in the intervention and comparison group hospitals using a difference-in-difference estimator. In addition, the investigators will conduct interviews with representatives from intervention hospitals to assess the extent to which ICAN hospitals implemented the CoC standards of cancer care.

DETAILED DESCRIPTION:
Intervention: The investigators received letters of support from hospitals, and those who direct the cancer center staff have expressed their willingness to participate on behalf of their staff. This is a health-system-level intervention, designed as single-arm intervention trial, where five participating hospitals will be offered support in the areas of training and education, cancer data collection and reporting, quality improvement and clinical peer-to-peer support.

The ICAN intervention was developed through implementation science processes as an adaptation of the Markey Cancer Center Affiliate Network (MCCAN) with retention of identified core functions. Each hospital in the intervention arm has undergone interviews about their current cancer program needs and offerings. From the information gathered through these meetings, the investigators established baseline understandings of cancer centers and their services. Through these meetings, the investigators elicited program goals, challenges, and readiness for change within their cancer services. Prior to starting the ICAN intervention, the cancer centers will be provided a documentation specifying current status for meeting CoC accreditation standards, gaps identified, suggestions and resources for the next steps to meet goals, and progress toward fulfilling CoC accreditation standards. Through the intervention, each of the five hospitals will be offered support, expertise, and resources necessary to facilitate hospitals in achieving the standards set forth by the American College of Surgeons Commission on Cancer. Support will be offered in the form of education and training regarding the standards and provision of cancer services, regular in-person and zoom check-ins with hospital stakeholders to evaluate progress, and provision of documentation and educational resources regarding standard requirements. The specific intervention actions will be tailored to the needs identified for each hospital or health system based on particular standards they currently do not meet and choose to work toward.

4 years from the start of the intervention, the investigators will use Iowa Cancer Registry data to evaluate the success of the intervention by comparing rates of compliance with pre- and post-intervention treatment-related quality measures in target and control hospitals using a difference-in-difference estimator. The rural hospitals in Iowa that serve the most rural cancer patients (all care for >100 newly diagnosed cancer patients per year) and have never been accredited by the CoC were chosen for intervention targets. The remainder of rural hospitals that care for >100 newly diagnosed cancer patients per year (n=4) were chosen as a comparison group. They were not contacted, as they will not be providing us with any data. Rather, the investigators will use data routinely collected by the Iowa Cancer Registry to compare aggregate compliance with quality measures for cancer care between the hospitals included in the intervention and hospitals that were not.

These variables needed to compute compliance with quality measures by hospital are routinely collected by the Iowa Cancer Registry from all hospitals in Iowa as part of routine public health surveillance. The investigators will only be using data provided to us by the Iowa Cancer Registry to calculate these measures for both intervention and control hospitals and will not be accessing medical record data from the intervention or control hospitals.

Interviews: Subjects from intervention hospitals will be asked to reply to the recruitment email and provide times over the subsequent two weeks that would for them to participate in a one-time audio/video-recorded telephone interview which will take approximately 30-45 minutes. Subjects will be asked prior to recording whether recording is permitted. If permitted, the interview will be recorded on zoom and converted to an audio file using UI (University of Iowa)-Capture. The recordings will be used to audio-transcribe the interview so that they transcript can be used in qualitative data-analysis. Only members of the research team will have access to the recordings. The audio-transcriptions will be done using the web-based service Rev.com. The recordings will be destroyed on completion of the data-analysis. The interview will include questions about the culture, structure, changes and current processes at their hospital for providing cancer care and the impact of the intervention. They will be mailed a $50 check in appreciation of their time after the interview has been conducted. There will be no additional follow-up to the interviews.

ELIGIBILITY:
Inclusion Criteria:

* Administrators, clinicians, and data monitoring staff who help provide cancer related care at one of the four hospitals that have been included in our study.

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance with CoC quality of cancer care measures: Hormone therapy (HT) | 36 months post implementation of intervention
  primary quality measure for breast cancer: percent of patients receiving tamoxifen or 3rd gen aromatase inhibitor within 1 year of diagnosis for women with T1cN0M0 or stage IB-III hormone receptor-positive cancer
Compliance with CoC quality of cancer care measures: 12 regional lymph nodes (12RLN) | 36 months post implementation of intervention
  primary quality measure for colon cancer: percent of patients having >12 regional lymph nodes removed and examined

SECONDARY OUTCOMES:
Compliance with CoC quality of cancer care measures: Breast conserving surgery radiation therapy (BCSRT) | 36 months post implementation of intervention
  percent of patients receiving radiation within 1 year of diagnosis for women <70 years old receiving breast conserving surgery for breast cancer
Compliance with CoC quality of cancer care measures: Multi-agent chemotherapy (MAC) | 36 months post implementation of intervention
  percent of patients receiving combination chemomotherapy within 4 months of diagnosis for women <70 years old with T1cN0M0 or stage IB-III hormone receptor-negative breast cancer
Compliance with CoC quality of cancer care measures: Adjuvant chemotherapy (ACT) | 36 months post implementation of intervention
  percent of patients receiving adjuvant chemotherapy within 4 months of diagnosis for patients <80 years old with AJCC Stage III (lymph node positive) colon cancer
Percentage of CoC evidence-based standards of cancer care implemented | 36 months post implementation of intervention
  Number and percentage of the 38 evidence-based CoC standards being met by each hospital

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroeder MC, Birken SA, Lizarraga IM, Kirk MA, Wagi CR, Engelbart JM, Johnson EC, Wahlen MM, Seaman AT, Charlton ME. Application of MODIFI to the adaptation of a complex, multilevel intervention to enhance access to high-quality cancer services in rural cancer hospitals. Implement Sci Commun. 2025 Oct 16;6(1):105. doi: 10.1186/s43058-025-00805-x. PMID 41102855